CLINICAL TRIAL: NCT03703531
Title: Effect of Duration of EMS Teams' Arrival on CPR Survival in Istria County, Croatia, 2011.-2017.
Brief Title: Istria County CPR Survival 2011-2017
Status: Completed | Type: Observational
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Andrej Šribar, Specialist in anesthesiology and intensive care medicine, Principal Investigator, University Hospital Dubrava
Other Study IDs: IstriaCPR
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cardiopulmonary Resuscitation
MeSH Terms: interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients resuscitated in Istria county: Cardiopulmonary resuscitation performed for OHCA
  Interventions: Procedure: Cardiopulmonary resuscitation

INTERVENTIONS:
Procedure: Cardiopulmonary resuscitation — CPR performed because of out-of-hospital cardiac arrest

SUMMARY:
Analysis of factors that influence CPR survival of 1440 patients that were resuscitated in Istria County, Croatia between 2011-2017.

DETAILED DESCRIPTION:
Survival status, duration to EMS arrival, level of education of initial CPR provider, initial monitored rhythm, cause of cardiac arrest, age, gender and time of year will be recorded and analyzed to determine which factors influence CPR survival.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients that were resuscitated in Istria county because of out of hospital cardiac arrest (OHCA)

Exclusion Criteria:

* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients resuscitated in the 2011-2017 time frame in Istria county, Croatia
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Survival status | At hospital admission
  Documented as electrocardiographic and hemodynamic evidence of return of spontaneous circulation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Dubrava, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No